CLINICAL TRIAL: NCT01754051
Title: VOLCAN: A Volumetric Coiling in Aneurysm Registry of the Penumbra Coil 400TM System
Brief Title: A Volumetric Coiling in Aneurysm Registry of the Penumbra Coil 400TM System
Acronym: VOLCAN
Status: Completed | Type: Observational
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP 4818; CLP 4818 (Other: Penumbra Inc)
Record Dates: First submitted 2012-12-17; First posted 2012-12-21 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Intracranial Aneurysms
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment by the PC 400 coils: Patients enrolled in this study must be those treated according to the cleared indication for the PC 400 System in the Instructions for Use.
  Interventions: Device: PC 400 coils

INTERVENTIONS:
Device: PC 400 coils

SUMMARY:
This study is a prospective, multi-center registry of patients with intracranial aneurysms who are treated by the PC 400 System. Data for each patient are collected up to 12 ± 3 months post-procedure for the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Intracranial aneurysms >2mm, ruptured or unruptured

Exclusion Criteria:

* Fusiform aneurysms
* Dissecting aneurysms
* Aneurysms associated with brain AVMs
* Multiple aneurysms
* Re-treated aneurysms
* Patients in whom endovascular embolization therapies other than PC 400 System are used will be excluded from this study. However, adjunctive use of balloon and stent are acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 200 patients with intracranial aneurysms treated by the PC 400 System at up to 20 centers will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-01; Primary Completion 2017-10-03 (Actual); Study Completion 2017-10-03 (Actual)

PRIMARY OUTCOMES:
Packing density with the number of coils implanted | During the procedure
Time of fluoroscopic exposure | During the procedure
Procedural device-related serious adverse events at immediate post-procedure | During the procedure
Quality of aneurysm occlusion post-operatively and at 12±3 months post-procedure based on the Raymond Scale | At 1 year post-procedure

SECONDARY OUTCOMES:
Acute occlusion of the aneurysm sac at immediate post-procedure | At immediate post-procedure
Adverse events occurring during the procedure and in the 30±7 days following the treatment. | During and at 30 days post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jérôme Berge, MD, Principal Investigator — CHU Pellegrin - Bordeaux
Locations (1):
- CHU Pellegrin, Bordeaux, France